CLINICAL TRIAL: NCT06687759
Title: A Phase 1 Study to Evaluate the Absorption, Distribution, Metabolism, and Excretion of [14C]MK-1084 in Healthy Adult Participants
Brief Title: A Study of MK-1084 Human Absorption, Distribution, Metabolism, and Excretion in Healthy Adult Participants (MK-1084-006)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1084-006; MK-1084-006 (Other: MSD)
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carbon-14 radiolabeled [14C] MK-1084 (Experimental): Participants receive single oral dose of MK-1084 on Day 1.
  Interventions: Drug: [14C]MK-1084

INTERVENTIONS:
Drug: [14C]MK-1084 — Oral administration

SUMMARY:
The purpose of this study is to learn what happens to MK-1084 in a healthy person's body over time and how it is cleared from the body.

ELIGIBILITY:
Inclusion Criteria:

Key inclusion criteria include but are not limited to the following:

* Is in good health based on medical history, physical examination,vital signs measurements, and electrocardiogram (ECG)s performed before randomization.
* Has a body mass index (BMI) 18 to 32 kg/m2, inclusive, at screening

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Has a history of cancer.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of plasma MK-1084 | Predose and at designated timepoints up to Day 15
  Bood samples will be collected to determine the AUC0-inf of MK-1084 in plasma.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of plasma MK-1084 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the AUC0-last of MK-1084 in plasma.
Area Under the Concentration-Time Curve from 0 to 24 hours (AUC0-24) of plasma MK-1084 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the AUC0-24 of plasma MK-1084 in plasma.
Maximum Concentration (Cmax) of plasma MK-1084 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the Cmax of MK-1084 in plasma.
Concentration at 24 hours postdose (C24) of plasma MK-1084 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the C24 of MK-1084 in plasma.
Time to Reach Maximum Concentration (Tmax) of plasma MK-1084 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the Tmax of MK-1084 in plasma.
Apparent Half Life (t½) of plasma MK-1084 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the t1/2 of MK-1084 in plasma.
Apparent Total Clearance (CL/F) of plasma MK-1084 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the CL/F of MK-1084 in plasma.
Apparent Volume of Distribution during the Terminal Elimination Phase (Vz/F) of plasma MK-1084 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the Vz/F of MK-1084 in plasma.
AUC0-inf/Total Radioactivity Ratio of plasma MK-1084 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the AUC0-inf/Total Radioactivity Ratio of MK-1084 in plasma.
Amount Excreted in the Urine (Aeu) of MK-1084 | Predose and at designated timepoints up to Day 15
  Urine samples will be collected to determine the Aeu of MK-1084
Cumulative Aeu of MK-1084 | Predose and at designated timepoints up to Day 15
  Urine samples will be collected to determine the cumulative Ae of MK-1084.
Percentage Excreted in the Urine (feu) of MK-1084 | Predose and at designated timepoints up to Day 15
  Urine samples will be collected to determine the feu of MK-1084.
Cumulative feu of MK-1084 | Predose and at designated timepoints up to Day 15
  Urine samples will be collected to determine the cumulative feu of MK-1084.
Amount Excreted in the Feces (Aef) of MK-1084 | Predose and at designated timepoints up to Day 15
  Feces samples will be collected to determine the Aef of MK-1084.
Cumulative Aef of MK-1084 | Predose and at designated timepoints up to Day 15
  Feces samples will be collected to determine the cumulative Aef of MK-1084.
Percentage Excreted in the Feces (fef) of MK-1084 | Predose and at designated timepoints up to Day 15
  Feces samples will be collected to determine the fef of MK-1084.
Cumulative fef of MK-1084 | Predose and at designated timepoints up to Day 15
  Feces samples will be collected to determine the cumulative fef of MK-1084.
Metabolites in Plasma of MK-1084 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the metabolites of MK-1084.
Metabolites in Urine of MK-1084 | Predose and at designated timepoints up to Day 15
  Urine samples will be collected to determine the metabolites of MK-1084.
Metabolites in Feces of MK-1084 | Predose and at designated timepoints up to Day 15
  Feces samples will be collected to determine the metabolites of MK-1084.

SECONDARY OUTCOMES:
Number of Participants Experiencing an Adverse Event (AE) | Up to ~ 28 days
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study treatment. For each arm, the number of participants experiencing an AE will be assessed.
Number of Participants Discontinuing Study Treatment due to an AE | Up to ~ 28 days
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study treatment. For each arm, the number of participants experiencing an AE will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Fortea CRU Madison (Site 0001), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/